CLINICAL TRIAL: NCT02525159
Title: Effectiveness of DIM Supplements to Increase 2-OHE1/16 Ratio in Premenopausal Mexican Women With Risk of Breast Cancer
Brief Title: Effectiveness of DIM Supplements to Increase 2-OHE1/16 Ratio
Acronym: EDIMI216OHE1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, Estela Ytelina Godínez Martínez, Researcher in Medical Sciences B, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SDEI.PTID.05.3(CM)
Record Dates: First submitted 2015-07-29; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
Keywords: 3,3'-diindolylmethane; premenopause; 2-hydroxyestrone
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DIM pills (Active Comparator): 75 mg of 3,3´-diindolylmethane (DIM) once a day for 30 days
  Interventions: Dietary Supplement: DIM pills
- Placebo pills (Placebo Comparator): 2 pills once a day for 30 days
  Interventions: Other: Placebo Pill

INTERVENTIONS:
Dietary Supplement: DIM pills — Two pills of BioResponse DIM® 150 are equal to 75 mg of DIM pure
  Other Names: BioResponse DIM® 150
  Arms: DIM pills
Other: Placebo Pill — Placebo pills, proportionate by the same provider, vials and pills were the same size, shape and material containing the DIM pills
  Arms: Placebo pills

SUMMARY:
Breast cancer is a public health problem in Mexico and its incidence rises when the woman is still premenopausal. Estrogen metabolism has been linked to breast cancer. Several studies reported that high concentrations of 2 hydroxyestrone (2OHE1) in urine have a protective effect for this neoplasia, whereas high concentrations of 16 alpha-hydroxyestrone (16αOHE1) in urine have the opposite effect, further has been reported that women with a ratio of estrogen metabolites 2OHE1:16αOHE1 in urine (REMU) less than 0.9, have ten times the risk of developing Breast Cancer than those women with an RMEU equal or more than 0.9. Other studies have showed that the active compounds of cruciferous vegetables, indole-3-carbinol (I3C) and its dimer, 3'3'diindolylmethane (DIM) induce benign pathway of metabolism of estrogens producing 2OHE1. Several studies, evaluate the pharmacokinetics and effect of I3C supplementation, finding that 300 to 600 mg of this compound are well tolerated and able to promote formation of 2OHE1 in women when supplemented for one month. In the case of DIM, only a pilot study has explored its effect in postmenopausal women with personal history of breast cancer in early stages, reporting an increase in the concentrations of 2OHE1. The purpose of this study was to evaluate the effectiveness of supplementation with DIM to increase urinary RMEU in premenopausal women at risk of Breast Cancer (RMEU less than 0.9). A clinical, randomized, double-blind study was performed with women attending on the urogynecology service of Institute National of Perinatology. Subjects were premenopausal women over 34 years who were healthy. The inclusion criteria's was had a RMEU less than 0.9 and were excluded for any medical condition, medication, or dietary or lifestyle habit that might interfere with estrogen metabolism. Patients were randomly assigned to one of two groups: one received orally at a daily dose of 75 mg of DIM for a period of 30 days and other group received orally at a daily placebo for a period of 30 days. All urine samples were collected from the women before DIM or placebo ingestion, after 30 days of DIM or placebo ingestion and finally after another 30 days once suspended supplementation. Analysis of the 2OHE1 and 16αOHE1 were determined using a commercially kit ESTRAMET™. The change in metabolites median concentrations and RMEU was assessed through the Wilcoxon test and these differences between groups through U Mann-Whitney test.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effectiveness of supplementation with 3,3´-Diindolylmethane (DIM) to increase the urinary ratio of estrogen metabolites 2OHE1:16alphaOHE1 (RMEU) in women at risk of breast cancer to contribute to generate a tool of early prevention of this disease.

Activities for detect women with REMU less than 0.9:

Check every day in the Institute National of Perinatology urogynecology service, clinical records of the women who attending consultations in order to verify the inclusion and exclusion criteria.

Interviewing these women to corroborate the inclusion and exclusion criteria. Quantify the concentrations of metabolites of estrogens in the urine for detect the presence of REMU less than 0.9.

Provide result and invite women who present REMU less than 0.9 to participate in the project of supplementation with DIM.

When women had a REMU equal or greater than 0.9, provide result and dietary guidance focused on maintaining BMI in normal range (19.0-24.9) or decrease (BMI more than or equal to 25) weight and the increase in the consumption of fruits and vegetables.

Activities for women inclusion in the study of DIM supplementation:

Once explained the study to the patients, women who met the criteria for inclusion were cited to provide an informed consent letter mentioning them that they had the freedom to clarify any doubt that might arise.

Once the woman read out the letter, understood it and agreed to participate, the signing of this was requested.

On the same date that each woman has signed the letter, another appointment was scheduled between day 12 and 15 of the menstrual cycle for the following assessments:

Personal data: Name, date of birth, address, phone, marital status and occupation.

Socioeconomic: With the criteria of the Mexican Association of Agencies of Market and Opinion based 2005

Complete clinical history that included:

Family history of chronic diseases included breast cancer, personal history of diseases and use medication, personal risk factors of breast cancer, type, frequency and duration of physical activity.

Nutrition: Whereas both anthropometric indicators (weight, height and perimeter wrist, waist and hip), body composition (% of body fat and lean mass by the method of displacement of air) and diet (24-hour recall, frequency of consumption of cruciferous vegetables in the last year and use of supplements). The measurements of anthropometric indicators were made using the LOHMAN technique. The information was processed with the NUTRIKCAL system that is standardized for foods commonly consumed in Mexico.

First morning urine. First morning urine with a difference no less than eight hours of previous urine.

Once urine samples were received, added them, for conservation, 0.1 g of ascorbic acid per 10 mL of urine, and stored at -70°C until it´s quantification.

For the analysis of the metabolites 2OHE1 and 16αOHE1, was used a competitive solid phase enzyme immunoassay method, using the commercial kit ESTRAMET™ 2/16 (Immune Care Corporation, Bethlehem, MI. USA), which was validated by the manufacturer by gas chromatography and mass spectrometry. The analysis was performed according to the manufacturer's instructions; briefly: the urine sample was hydrolyzed with an enzyme beta glucuronidase and sulfatase activities. The free urinary metabolites, joined to monoclonal antibodies conjugated with alkaline phosphatase. The quantification of metabolites 2OHE1 and 16αOHE1 were performed in triplicate and the reproducibility of this method has already been reported by our team in a study. For each of the determinations of the RMEU were reference curves, achieving a 97% of accuracy.

Adherence and side effects. In the first assessment is gave women a calendar to daily record consumption or omission of the supplement (active compound or placebo) as well as a series of side effects in order to assess the adherence and safety of supplement. This included side effects that had already been reported in other studies with DIM and I3C. In addition requested participants return the supplements vial to subsequently make the count of pills that were left over.

Sample size.

To estimate the sample size it was considered the following:

Two sets of comparison (Placebo and 75mg DIM). According to literature and hoping to find a difference of .48 in the average of RMEU of the group of supplementation relative to the placebo group.

Other studies have reported a standard deviation of .77 on the RMEU. Calculated with an alpha of 0.05 and a power of 80%. Approximately 31 women are required by group plus 10% to replace losses in the follow-up, which gives an approximate total of 35 women per group.

Statistical Analysis. The statistical analysis of data was carried out in the following way: the differences between baseline characteristics was performed using the student T test for parametric variables with normal distribution, U Mann-Whitney for those who did not have a normal distribution and X2 for the nonparametric. The change of estrogen metabolites and RMEU in each group was evaluated using the Wilcoxon test and the comparison of the effect between groups, the values of concentrations of the metabolites of estrogen and the RMEU as well as their differences, was carried out by means of the test U Mann-Whitney.

Masking. A stranger to the study researcher, received and coded vials containing the DIM supplement and placebo, recording the code in a role that was kept in an envelope that was opened at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman
* Not pregnant or planning to become pregnant
* That are not nursing
* Nonsmokers
* No alcohol addiction
* Regular menstrual cycles
* 2-hydroxyestrone /16 urinary ratio less or equal to 0.9

Exclusion Criteria:

* Take drugs that interfere with estrogen metabolism like hormonal contraceptives , cimetidine , antidepressants, thyroxine , supplements of n-3 fatty acids or soy
* Endocrine or liver disease
* Pregnancy

Ages: 35 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in ratio of estrogen metabolites 2OHE1:16αOHE1 in urine (REMU) | At day 0, at day 30 after the supplementation of DIM or placebo and 30 days after the end of the suplementation of DIM or placebo to evaluate the permanence of the response

SECONDARY OUTCOMES:
Adherence | Dialy, after the day 0 until the end of the supplementation of DIM or placebo (day 30)
  A schedule was provided to the patients to record the daily intake of the supplement DIM/placebo
Presence of Side Effects | At day 0 and 30 days after the supplementation of DIM or placebo
  A schedule was provided to the patients to record daily the presence of side effects that have been reported in other studies such as diarrhea, nausea , vomiting , headache and flatulence.

OTHER OUTCOMES:
Prolonged use of hormonal contraceptives | At day 0
  Use for five years or more
Late pregnancy or nulliparity | At day 0
  First pregnancy after 35 years or no living children
Age | At day 0
Family history of breast cancer | At day 0
  Have at least one first-degree or second degree family, who has had or have the disease
Early menarche | At day 0
  Age at first period at twelve or more
Body Mass Index (IMC) | At day 0, at day 30 after the suplementation of DIM or placebo and 30 days after the end of the suplementation of DIM or placebo
% of body fat | At day 0, at day 30 after the suplementation of DIM or placebo and 30 days after the end of the suplementation of DIM or placebo
Waist perimeter | At day 0, at day 30 after the suplementation of DIM or placebo and 30 days after the end of the suplementation of DIM or placebo
Physical activity | At day 0, at day 30 after the suplementation of DIM or placebo and 30 days after the end of the suplementation of DIM or placebo
  More than 150 minutes per week
Socioeconomic level | At day 0
  According to the committee of socioeconomic levels of the Mexican Association of Market Research Agencies and Public Opinion (AMAI)
Consumption of cruciferous vegetables | At day 0, at day 30 after the suplementation of DIM or placebo and 30 days after the end of the suplementation of DIM or placebo
  Number of portions per day (1 cup raw or 1/2 cup cooked) of any cruciferous vegetables

REFERENCES:
- [Background] Falk RT, Rossi SC, Fears TR, Sepkovic DW, Migella A, Adlercreutz H, Donaldson J, Bradlow HL, Ziegler RG. A new ELISA kit for measuring urinary 2-hydroxyestrone, 16alpha-hydroxyestrone, and their ratio: reproducibility, validity, and assay performance after freeze-thaw cycling and preservation by boric acid. Cancer Epidemiol Biomarkers Prev. 2000 Jan;9(1):81-7. PMID 10667467
- [Background] Godinez Martinez EY, Santillan Ballesteros R, Lemus Bravo AE, Samano R, Tolentino Dolores M, Rodriguez Ventura AL, Juarez Gonzalez AR. [Determination of 2-hydroxyestrone /16alpha-hydroxyestrone ratio in urine of Mexican women as a risk indicator for breast cancer and its relationship with other risk factors]. Nutr Hosp. 2014 Oct 25;31(2):835-40. doi: 10.3305/nh.2015.31.2.8172. Spanish. PMID 25617571
- [Background] Reed GA, Peterson KS, Smith HJ, Gray JC, Sullivan DK, Mayo MS, Crowell JA, Hurwitz A. A phase I study of indole-3-carbinol in women: tolerability and effects. Cancer Epidemiol Biomarkers Prev. 2005 Aug;14(8):1953-60. doi: 10.1158/1055-9965.EPI-05-0121. PMID 16103443
- [Background] Dalessandri KM, Firestone GL, Fitch MD, Bradlow HL, Bjeldanes LF. Pilot study: effect of 3,3'-diindolylmethane supplements on urinary hormone metabolites in postmenopausal women with a history of early-stage breast cancer. Nutr Cancer. 2004;50(2):161-7. doi: 10.1207/s15327914nc5002_5. PMID 15623462
- [Background] Wong GY, Bradlow L, Sepkovic D, Mehl S, Mailman J, Osborne MP. Dose-ranging study of indole-3-carbinol for breast cancer prevention. J Cell Biochem Suppl. 1997;28-29:111-6. doi: 10.1002/(sici)1097-4644(1997)28/29+3.0.co;2-k. PMID 9589355
- See also: Association of Market Research Agencies and Public Opinion 2005 — http://www.amai.org
- See also: Inmune Care Corporation. USA. — http://www.immunacare.com/proto-col.htm
- See also: Studies with the ESTRAMET™ 2/16 kit — http://www.immunacare.com/studies.htm